CLINICAL TRIAL: NCT00153686
Title: Capsule Endoscopy or Mesenteric Angiogram in Patients With Overt Gastrointestinal Bleeding of Obscure Origin: A Randomized Study
Brief Title: Capsule Endoscopy or Mesenteric Angiogram in Patients With Overt Gastrointestinal Bleeding (GIB) of Obscure Origin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: WK Leung, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CE_Ang
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-05-13 (Estimated); Status verified 2008-05

CONDITIONS: Gastrointestinal Hemorrhage
Keywords: Capsule Endoscopy; Mesenteric angiogram
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capsule Endoscopy (Experimental): Capsule Endoscopy examination of small intestine
  Interventions: Procedure: capsule endoscopy
- Mesenteric Angiogram (Other): Mesenteric Angiogram of the small intestine
  Interventions: Procedure: Mesenteric Angiogram

INTERVENTIONS:
Procedure: capsule endoscopy — capsule endoscopy of small intestine
  Arms: Capsule Endoscopy
Procedure: Mesenteric Angiogram — Mesenteric Angiogram
  Arms: Mesenteric Angiogram

SUMMARY:
To compare the diagnostic yield of mesenteric angiogram with CE in patients with active obscure GIB.

DETAILED DESCRIPTION:
Gastrointestinal bleeding (GIB) of obscure origin is a common conditions resulting in recurrent hospitalization and extensive investigations. Mesenteric angiogram is one of the standard radiological investigations for GIB of obscure origin, and its diagnostic yield ranged from 40-80%. Capsule endoscopy (CE) is a newly available investigation for small bowel examination, especially in bleeding of obscure origin. The diagnostic yield is particularly high in patients with ongoing bleeding. This is a prospective randomized study to compare the diagnostic yield of mesenteric angiogram with CE in patients with overt GIB of obscure origin. The results will help to define the optimal management strategy for this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to PWH medical or surgical wards with melena or hematochezia in whom OGD and colonoscopy fail to identify site of bleeding.
* Normal or non-diagnostic OGD and colonoscopy
* Informed consent
* Patients presented with shock will be resuscitated for urgent endoscopy

Exclusion Criteria:

* Patients remained in shock despite resuscitation.
* Moribund patients
* Terminal malignancy
* Presence of pacemaker or ICD
* Suspected or confirmed intestinal obstruction
* Swallowing difficulties
* Renal failure that preclude angiographic examination
* Pregnancy
* Age <18
* Refused consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2005-06; Primary Completion 2007-11 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of CE and mesenteric angiogram as the primary investigation after negative EGD and colonoscopy. | 12 months

SECONDARY OUTCOMES:
Percentage of patients with definitive diagnoses achieved;Length of stay (days) ;Transfusion requirements;No. of additional investigations (endoscopies, radiological investigation, CE etc);No. of patients requiring surgery ;12-month rebleeding rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wai K Leung, MD, Principal Investigator — CUHK
Locations (1):
- Endoscopy Center, Prince of Wales Hospital, Hong Kong(SAR), China